CLINICAL TRIAL: NCT01319799
Title: Microembolic Signals and Cerebrospinal Fluid Markers of Neuronal Damage After Surgical Aortic Valve
Brief Title: Microembolic Signals and Cerebrospinal Fluid Markers of Neuronal Damage After Surgical Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bjorn Reinsfelt, Consultant MD, PhD,Cardiothoracic Anaesthesia, Sahlgrenska University Hospital
Other Study IDs: Dnr112-09
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Aortic Stenosis
Keywords: Embolism; Nervous system; Aorta; Valves; Ultrasonics
MeSH Terms: conditions — Aortic Valve Stenosis; Embolism; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid levels of S100B, NSE , Tau and albumin detected by elctrochemoluminescence immunoassay.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical aortic valve replacement: Single observational study. Count of microembolic signals during open heart surgery and measurement of properative vs postoperative levels of markers in cerebrospinal fluid of neuronal damge.
  Interventions: Other: Open heart surgery

INTERVENTIONS:
Other: Open heart surgery — TCD count of microembolic signals during surgical aortic valve replacement

SUMMARY:
The use of MRI have shown that the incidence of postoperative cerebral lesions due to cerebral embolization is high (1). Nonetheless the extent of postoperative neurological dysfunction is only a fraction of the actual amount of new postoperative changes detected on MRI. Transcranial Doppler (TCD) has shown the occurrence of extensive microembolic signals in intracerebral arteries during open heart procedures (2). The clinical significance of cerebral microemboli is not clear (3-5). The use of serological markers to assess cerebral injury after open cardiac surgery is difficult to interpret. The levels of markers seems to be contaminated from extracerebral sources (6). In order assess the release of markers of neuronal damage after open aortic valve surgery the investigators intend to examine the levels of S-100B, NSE and Tau in cerebrospinal fluid (CSF) by comparing the levels preoperative with the levels one day after surgery. Furthermore the investigators will determine the total amount of cerebral microembolic signals during the surgical procedure by means of TCD. The investigators will statistically test if there is any correlation between the increase in cerebrospinal fluid levels of S-100B,NSE and Tau and the cerebral embolic load.

DETAILED DESCRIPTION:
Patients and clinical procedures 10 patients scheduled for open aortic valve surgery at our institution will be included into this prospective, observational study. The Human Ethics Committee of the University of Gothenburg, approved the study protocol. The day before surgery a lumbar puncture at level L3-4 will be performed using a 27G Whitacre needle. A sample of 2.5 ml of cerebrospinal fluid will be taken for analysis of S-100B, NSE, Tau and albumin.

On arrival at OR, standard perioperative monitoring will be established, including an Auditory Evoked Potential (AEP) monitor for anaesthetic depth measurements (AEP Monitor/2, Danmeter, Odense, Denmark) and radial arterial and central venous lines. General anaesthesia is induced with propofol 0.5-1 mg/kg and fentanyl 10 μg/kg. Tracheal intubation will be facilitated using atracurium 0,5 mg/kg. Sevoflurane is used to maintain an anaesthetic depth adjusted to an AAI index of 15-30 as recorded by the AEP monitor. Hemodynamic stability will be obtained by the use of colloidal solution administration, guided by the use of intra-operative transesophageal echocardiography, and norephineprine to maintain a mean arterial pressure above 75 mmHg-Also during CPB. A lumbar puncture will be repeated the first postoperative day repeating the measurement of markers in CSF A certified cardiologist or anaesthesiologist assess focal neurological impairment before and within 24 hours after the procedure.

Transcranial Doppler (TCD) By TCD the right medial cerebral artery (RMCA) will be insonated by the transtemporal approach at a depth of approximately 50 mm using standard criteria. The investigators use a 2 MHz power M-mode TCD monitor (ST3 ©, Spencer Technologies Seattle, WA), with the probe fixed in position using a head frame. The Doppler signals will be continuously monitored and saved to monitor hard drive. Two physicians independently evaluate the TCD data files offline, and identify microembolic signals (MES) using criteria for counting emboli signals on spectral and PMD TCD.

Statistical Analysis: Descriptive statistics and tests of normality for continuos data Correlation analysis; Total cerebral embolic load vs. increase of CSF level S-100B/ NSE/Tau.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis aortic stenosis eligible for surgical treatment

Exclusion Criteria:

* Coagulopathy
* Regular Anticoagulation therapy
* Carotid stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elective surgical aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Erik Ricksten, Professor, Study Director — Sahlgrenska University Hospital,Thoracic Anesthesia & Intensive Care
Locations (1):
- Department of Thoracic Anaesthesia & Intensive Care,Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stolz E, Gerriets T, Kluge A, Klovekorn WP, Kaps M, Bachmann G. Diffusion-weighted magnetic resonance imaging and neurobiochemical markers after aortic valve replacement: implications for future neuroprotective trials? Stroke. 2004 Apr;35(4):888-92. doi: 10.1161/01.STR.0000120306.82787.5A. Epub 2004 Feb 19. PMID 14976326
- [Background] Abu-Omar Y, Balacumaraswami L, Pigott DW, Matthews PM, Taggart DP. Solid and gaseous cerebral microembolization during off-pump, on-pump, and open cardiac surgery procedures. J Thorac Cardiovasc Surg. 2004 Jun;127(6):1759-65. doi: 10.1016/j.jtcvs.2003.09.048. PMID 15173734
- [Background] Kruis RW, Vlasveld FA, Van Dijk D. The (un)importance of cerebral microemboli. Semin Cardiothorac Vasc Anesth. 2010 Jun;14(2):111-8. doi: 10.1177/1089253210370903. PMID 20478951
- [Background] van Dijk D, Kalkman CJ. Why are cerebral microemboli not associated with cognitive decline? Anesth Analg. 2009 Oct;109(4):1006-8. doi: 10.1213/ANE.0b013e3181b5af06. No abstract available. PMID 19762723
- [Background] Martin KK, Wigginton JB, Babikian VL, Pochay VE, Crittenden MD, Rudolph JL. Intraoperative cerebral high-intensity transient signals and postoperative cognitive function: a systematic review. Am J Surg. 2009 Jan;197(1):55-63. doi: 10.1016/j.amjsurg.2007.12.060. Epub 2008 Aug 23. PMID 18723157
- [Background] Anderson RE, Hansson LO, Nilsson O, Liska J, Settergren G, Vaage J. Increase in serum S100A1-B and S100BB during cardiac surgery arises from extracerebral sources. Ann Thorac Surg. 2001 May;71(5):1512-7. doi: 10.1016/s0003-4975(01)02399-2. PMID 11383792

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Aortic Valve Replacement: Open heart surgery : TCD count of microembolic signals during surgical aortic valve replacement
Period: Overall Study
Arm/Group | Surgical Aortic Valve Replacement
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgical Aortic Valve Replacement
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Transcranial Doppler(TCD) Microembolic Signals During Surgical Aortic Valve Replacement Surgery
Description: Transcranial Doppler measurement of microembolic signals will be measured during the surgical procedure.Microembolic signals are detected by offline analysis of the Dopplerspectral analysis of the blood flow in the medial cerebral artery. Different intensities (dB),flow direction and time frame appearances in the Doppler spectral envelope is distinguishable for a neurosonolgist according to predefined criteria for an embolic signal-defined in previous litterature.The total amount of signals during one surgical procedure is counted. The appearance of microembolic signals related to specific procedures performed during cardiac surgery with cardiopulmonary bypass is noted. The exact time range is not possible to estimate in advance,due to the fact that each surgical procedure varies in time.The range of values for each individual patient, based on pilos, will vary from 50 to approximately 1500 embolic counts for one surgical procedure. A high value is negative for the patient.
Time Frame: (day 1) TCD will be performed from start of surgery till end of surgery-exact time cannot be stated in advance
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Surgical Aortic Valve Replacement
Number analyzed (Participants) | 10
units on a scale | 354 (79)

2. Secondary Outcome: Cerebrospinal Fluid(CSF) Levels of S-100B(Microgram/Liter)
Description: Differences in preoperative vs postoperative CSF levels of S-100B in microgram/Liter
  The assumption is that a cardiac open heart surgical procedure with cardiopulmonary bypass will influence the postoperative level of marker of neuronal cell damage in the central nerve system. An increase in the levels, compared to the preoperative values, indicates neuronal cell damage detectable in the CSF, namely the brains own extracellular fluid.
Time Frame: 24 Hours after Surgery
Measure: Mean (Standard Error); unit: microgram/Liter
Arm/Group | Surgical Aortic Valve Replacement
Number analyzed (Participants) | 10
microgram/Liter | 0.11 (0.02)

ADVERSE EVENTS:
Arm/Group | Surgical Aortic Valve Replacement
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
100 patients asked for participation; 10 accepted. Large outcome in descriptive study- Ended after 10 cases

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes